CLINICAL TRIAL: NCT05751122
Title: Effects of Dynamic Flex Cast With Neurodevelopmental Treatment on Gross Motor Functions in Children With Cerebral Palsy
Brief Title: Effects of Dynamic Flex Cast With Neurodevelopmental Treatment on Gross Motor Functions in Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Nafisa Gul
Record Dates: First submitted 2023-02-20; First posted 2023-03-02 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Cerebral Palsy
Keywords: Ankle joint; Cerebral Palsy; Spasticity; Dynamic cast
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dynamic flex cast with neurodevelopmental Group (Experimental): Dynamic flex cast with neurodevelopmental treatment
  Interventions: Other: Dynamic flex cast with neurodevelopmental treatment
- Rigid Ankle foot Orthosis with neurodevelopmental Group (Active Comparator): Rigid Ankle foot Orthosis with neurodevelopmental treatment
  Interventions: Other: Rigid Ankle foot Orthosis with neurodevelopmental treatment

INTERVENTIONS:
Other: Dynamic flex cast with neurodevelopmental treatment — Neurodevelopmental therapy in combination with dynamic flex cast to treat experimental group.
  Three times a week, 1 hour session per day.
  Dynamic flex casting is casting which manipulate bone alignment and maintains range of motion or sustained stretch. Casting will be changed weekly for 3 months.
  Neuro developmental approach is individualized treatment which is attuned to each child's specific problems, aims and goals.
  Key elements in NDT are: facilitation (using sensory inputs to improve motor performance), management of compensatory motor behavior, and an overall management strategy (a 24-hour interdisciplinary management approach) NDT involves task specific postures and movements.
  Arms: Dynamic flex cast with neurodevelopmental Group
Other: Rigid Ankle foot Orthosis with neurodevelopmental treatment — Rigid ankle foot orthosis will be applied to ankle joint at the start of intervention.
  Neurodevelopmental treatment will be applied to both groups with protocol; Three times a week, 1 hour session per day.
  Assessment on 1st day,6th week and 12th week
  Arms: Rigid Ankle foot Orthosis with neurodevelopmental Group

SUMMARY:
The study aims to determine the effects of dynamic flex cast with neurodevelopmental treatment on gross motor functions and gait in children with cerebral palsy.

DETAILED DESCRIPTION:
The study aims to determine the effects of dynamic flex cast with neurodevelopmental treatment on gross motor functions and gait in children with cerebral palsy. Combination of Dynamic flex cast with neurodevelopmental treatment will be a novel potential treatment to improve gross motor functions in cerebral palsy. We shall try to fill the gaps of previous studies. It will help in facilitating children to perform their activities, restoring normal ranges and treatment of spasticity in cerebral palsy.

ELIGIBILITY:
Inclusion Criteria:

* Children with cerebral palsy
* Age 3-8 years
* Spastic diplegic/ hemiplegic CP
* Ankle dorsiflexion 5-10 degrees
* GMFCS level 1-3
* Modified Ashworth's scale level 1+ - 3

Exclusion Criteria:

* Congenital foot deformities
* Cognitive impairments
* Secondary orthopedic, auditory and severe visual impairments
* Unwilling patients or parents
* Recent surgical interventions

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2023-02-25 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
Gross Motor Function Measure-88 | 12 weeks
  The original GMFM has 88 items each scored on a 4-point ordinal scale of 0 to 3, where 0 indicates that the child does not initiate the task; 1 indicates that the child initiates the task (completes < 10% activity); 2 indicates that the child partially completes the task (completes from 10 to 99% of activity); 3 indicates that the child completes the task (100%); and NT indicates that the child was not tested. The 88 items are grouped into five dimensions: 1) lying and rolling, 2) sitting, 3) crawling and kneeling, 4) standing, and 5) walking, running and jumping. Reliability with intraclass correlation coeffcient greater than .98 with 0.965--.994 95% confidence interval.
Clinical Gait Assessment Scale | 12 weeks
  It is used to assess gait deviation. Temporal distance factors including velocity, cadence, stride length, stride width will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Abrish Abbasi, MS-NMPT, Principal Investigator — Riphah International University
Locations (1):
- Chal foundation, Bacha Khan Medical Complex, Swābi, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No